CLINICAL TRIAL: NCT04333667
Title: Effectiveness of Mindfulness-based Internet Intervention Still Me: a Randomized Controlled Trial
Brief Title: Effectiveness of Mindfulness-based Internet Intervention Still Me
Acronym: Still-Me
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vilnius University (Other)
Collaborators: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Evaldas Kazlauskas, Professor, Vilnius University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-02-27/36
Record Dates: First submitted 2020-03-31; First posted 2020-04-03 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Post-traumatic Stress Disorder
Keywords: PTSD; mindfulness; efficacy; internet intervention
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated either to the intervention or control groups. The control group is a waiting list. The control group will participate in the intervention after it will be completed for the intervention group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group will get an 8-week mindfulness-based internet intervention.
  Interventions: Behavioral: Intervention group
- Control group (No Intervention): The waiting list will get no intervention while the intervention group is getting the intervention. The waiting list has the possibility to get an intervention after the intervention group finishes it.

INTERVENTIONS:
Behavioral: Intervention group — The intervention consists of 8 modules. Each week participants get access to a new module. Each module consists of psychoeducation and exercise parts. Most of the exercises are based on audio records. The content of the modules includes such themes as awareness and nonjudgement of senses, emotions, and thoughts. Participants can reach a psychologist on demand.
  Arms: Intervention group

SUMMARY:
The aim of the study is to assess the effectiveness of a mindfulness-based internet intervention for post-traumatic stress disorder symptoms.

DETAILED DESCRIPTION:
Intervention is going to take the form of a mindfulness-based internet intervention consisting of eight modules. The themes include awareness and nonjudgment of senses, emotions, and thoughts. These themes were chosen after considering topics that might be the most useful for individuals who experience post-traumatic disorder symptoms. Each module consists of psychoeducation and exercise (audio records mostly) parts. Psychologist can be reached on demand.

The effect of the intervention will be compared against a waiting list control group. Intervention is in Lithuanian.

ELIGIBILITY:
Inclusion Criteria:

* at least 18-years-old;
* understand Lithuanian;
* internet access and device for that;
* at least one traumatic event during lifetime;
* post-traumatic stress disorder symptoms.

Exclusion Criteria:

* an acute case of psychiatric care;
* interpersonal violence;
* alcohol / drug addiction;
* cannot participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2020-04-14 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change on International Trauma Questionnaire | Pre-treatment, after 8 weeks, 3 months post-treatment
  Changes on post-traumatic stress disorder are measured. International Trauma Questionanaire (ITQ, Cloitre et al., 2018) is a self-report measure and consists of 18 questions. All items are answered on a 5-point Likert scale that ranges from 0 (not at all) to 4 (extremely). Higher score indicates more pronounced symptoms.

SECONDARY OUTCOMES:
Change on Patient Health Questionnaire-9 | Pre-treatment, after 8 weeks, 3 months post-treatment
  Changes on depression symptoms are measured. Patient Health Questionnaire-9 (PHQ-9, Kroenke et al., 2001) is a self-report measure and consists of 9 questions. All items are answered on a 4-point Likert scale that ranges from 0 (not at all) to 3 (nearly every day). Higher score indicates more pronounced symptoms.
Change on General anxiety disorder | Pre-treatment, after 8 weeks, 3 months post-treatment
  Changes on anxiety symptoms are measured. General Anxiety disorder (GAD-7, Spitzer, Kroenke, Williams, & Löwe, 2006) is a self-report measure and consists of 7 items. All items are answered on a 4-point Likert scale that ranges from 0 (not at all) to 4 (nearly every day). Higher score indicates more pronounced symptoms.
Change on Adjustment disorder - New Module 8 | Pre-treatment, after 8 weeks, 3 months post-treatment
  Changes on adjustment disorder are measured. Adjustment disorder - New Module 8 (ADNM-8, Kazlauskas et al., 2018) is a self-report measure comprised of two parts: the stressor list, and the symptom list. The symptom list answers are answered on a 4-point Likert scale that ranges from 1 (never) to 4 (often).Higher score indicates more pronounced symptoms.
Change on Positive Mental Health Scale | Pre-treatment, after 8 weeks, 3 months post-treatment
  Chages on positive mental health are measured. Positive Mental Health Scale (PMH, Lukat et al., 2016) is a self-report measure and consists of 9 questions. All items are answered on a 4-point Likert scale that ranges from 0 (do not agree) to 3 (agree). Higher score indicates more pronounced positive mental health.
Change on Five Facet Mindfulness Questionnaire-Short form | Pre-treatment, after 8 weeks, 3 months post-treatment
  Changes on mindfulness skills are measured. Five Facet Mindfulness Questionnaire-Short form (FFMQ-SF, Bohlmeijer et al., 2011) is a self-report measure and consists of 24 items. All items are answered on a 4-point Likert scale that ranges from 1 (never or very rarely true) to 5 (very often or always true). Higher score indicates more pronounced mindfulness skills.

CONTACTS AND LOCATIONS:
Overall Officials: Evaldas Kazlauskas, Ph.D., Principal Investigator — Vilnius University
Locations (1):
- Vilnius University, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dumarkaite A, Truskauskaite-Kuneviciene I, Andersson G, Kazlauskas E. The Effects of Online Mindfulness-Based Intervention on Posttraumatic Stress Disorder and Complex Posttraumatic Stress Disorder Symptoms: A Randomized Controlled Trial With 3-Month Follow-Up. Front Psychiatry. 2022 Mar 30;13:799259. doi: 10.3389/fpsyt.2022.799259. eCollection 2022. PMID 35432020